CLINICAL TRIAL: NCT05406154
Title: A Multicenter Prospective Observational Study to Evaluate the Safety and Efficacy of Ibrutinib Combined With Bendamustine and Rituximab in Newly Diagnosed Mantle Cell Lymphoma Patients Who Aged > 65 Years
Brief Title: Ibrutinib Combined With Bendamustine and Rituximab in Newly Diagnosed Mantle Cell Lymphoma Patients Who Aged > 65 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Peking University First Hospital (Other); Beijing Tongren Hospital (Other); Beijing Hospital (Other Government); Beijing Tsinghua Changgeng Hospital (Other); China-Japan Friendship Hospital (Other); 307 Hospital of PLA (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Harbin Medical University (Other); Baotou Cancer Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Shanxi Province Cancer Hospital (Other); Beijing Naval General Hospital (Other); First Hospital of China Medical University (Other); Jilin Provincial Tumor Hospital (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021031
Record Dates: First submitted 2021-07-08; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-06

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: MCL; Ibrutinib; aged > 65 years
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a prospective observational clinical trial. A total of 19 research centers were involved in this study. Each site plans to enroll 2-3 patients, and a total of 60 patients will be enrolled. Patients who met the diagnosis of mantle cell lymphoma by histological examination, ECOG (Eastern Oncology Collaborative Group) score 0-2, age >65 years, expected survival of more than 3 months, and at least one measurable lesion were included in this observational clinical trial. In this study, clinical data of patients treated with R-B regimen combined with ibrutinib will be collected, including routine clinical laboratory tests, examinations, and molecular biological data, for efficacy assessment and survival analysis. The main evaluation indicators are the total effective rate of 2 and 6 cycles of alternating R-CHOP/R-DHAP combined with ibrutinib in the treatment of newly treated muff cell lymphoma patients. The 3-year progression-free survival (PFS) and overall survival (OS) of the patients will be assessed, and adverse events to treatment will be collected to evaluate the safety of ibrutinib in combination with untreated mask cell lymphoma.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is a B-cell lymphoma with unique histomorphology、immunophenotype and cytogenetic characteristics, accounting for 6% to 8% of non-Hodgkin's lymphoma, occurs in older men, with a median age of 68 years old, male: female is about 2 to 4:1, 80% of patients during the diagnosis is in progress, both indolent and aggressive lymphoma inert lymphoma incurable characteristic. The main clinical manifestations were lymph node and hepatosplenomegaly. Extranodal involvement is common, and the commonly involved sites include bone marrow, gastrointestinal tract, and Waldeyer'sring [1], t (11; 14) (q13; q32) Excessive expression in the Cyclin D1 nucleus caused by abnormalities is characteristic of MCL. In recent years, although the application of new drugs has made a lot of progress in the treatment of mantle cell lymphoma, the overall efficacy is not good, the vast majority of patients relapse after treatment, the median survival of 3-5 years, the lack of standard treatment regimens[2.3]. Blast-cell type and high-risk mantle cell lymphoma account for 10-15%, with higher clinical invasiveness and poorer prognosis.

For older patients with MCL, treatment regimens and objectives should be adjusted according to risk factors. Current studies have shown that both BR regimen (rituximab + bendamustine) and R-CHOP regimen can be used in elderly patients with MCL. Previously studies have shown that initial treatment indolent B cell lymphoma and mantle cell lymphoma, BR and R - CHOP plan randomized controlled studies show that BR scheme can significantly the patient's complete remission rate (40% vs 30%, P = 0.021) and progression-free survival (69.5 m vs. 31.2 m, P < 0.0001), and BR group 3-4 patients with leukopenia and incidence of infection were significantly reduced[4]. The phase III Ⅱ clinical trial showed that 57 MCL patients with a median age of 71 years were enrolled in the R-BAC500 regimen for 4-6 cycles. The results showed that the ORR of the patients was 96%, the CR rate was 93%, 51% of the patients achieved bone marrow MRD negative, the 2-year PFS rate was 81%, the OS rate was 85%, and the hematological adverse reactions were significantly reduced[5,6]Based on the above studies, BR-based treatment regimen has become the first-line treatment regimen for senile mantle cell lymphoma[7,8]. Recurrence of elderly set of cell lymphoma, face the same problem, 60% of cell lymphoma in patients with disease recurrence after first-line treatment, once the elderly patients with recurrence after treatment effect is poorer, so how to improve the elderly mantle cell lymphoma patients reponse depth, reduce disease relapse, has become an important treatment goal of mantle cell lymphoma.

Ibrutinib, as a BTK inhibitor, has shown significant efficacy in the treatment of mantle cell lymphoma, and has become an important choice in the treatment of mantle cell lymphoma[9] . The PCYC1104 clinical study showed that ibrutinib monotherapy was used to treat recurrent and refractory mantle cell lymphoma with a median follow-up of 15.3 months, with a CR21%, PR47%, ORR68%, and median PFS13.9 months[10,11]; Another randomized, open, multi-center phase III trial comparing ibrutinib to Temsirolimus monotherapy in relapsed and refractory mantle cell lymphoma showed a statistically significant difference in CR18.7%, PR53.2%, ORR72%and median PFS15.6 months compared with sirolimus monotherapy[12]. Based on these studies, ibrutinib is now an important treatment option for relapsed and refractory mantle cell lymphoma recommended by various guidelines. The significant efficacy of ibrutinib in the treatment of mantle cell lymphoma has been studied both at home and abroad. Ibrutinib is used for the treatment of elderly patients with mantle cell lymphoma at the initial treatment, and combined treatment with ibrutinib can achieve deep complete remission and reduce disease recurrence.The haematology annual report 2019, 50 cases treated first in elderly patients with sets of cell lymphoma with zlatan ibrahimovic for combined therapy with mabthera, continued until disease progression, oral CR60% after combined treatment, ORR98%, 81% patients achieve MRD negative, the study for ibrahimovic, combination therapy in the elderly set of cell lymphoma treated first provide treatment, has become an old set of cell lymphoma treated first important treatment options.

The retrospective analysis of 256 cases of Chinese patients with mantle cell lymphoma showed that the survival rate of Chinese patients with mantle cell lymphoma after initial treatment was 40.9%, Orrin 81.6%, 5-year PFS51.2% and 5-year OS58.4%, which were significantly lower than that of foreign patients with mantle cell lymphoma. Among them, the elderly patients aged over 65 years accounted for 33.2%. Compared with young patients, the elderly MCL had poor chemotherapy tolerance, and the complete remission rate and overall survival were significantly lower than those of young patients. Therefore, the initial treatment for elderly mantle cell lymphoma patients in the Chinese population needs to be further optimized. As a BTK inhibitor with the longest marketing history, ibrutinib has been widely used in the clinical treatment of mantle cell lymphoma and listed in NRDL.In clinical treatment, ibrutinib combined with BR regimen has been used for elderly patients, showing a good complete response rate and tolerable safety. In order to better collect the clinical data of ibrutinib combined with BR regimen and make a more scientific and accurate evaluation, the observational clinical study on the safety and efficacy of R-B regimen combined with ibrutinib in the initial treatment of mask cell lymphoma at the age of > age 65 was carried out in our center. This study was able to collect the ORR of 2 and 6 cycles of R-B combined with ibrutinib treatment in the Chinese population of elderly manusol cell lymphoma in the initial treatment, evaluate the survival indicators, and collect the adverse reactions during the treatment and the recurrence rate after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 65 years old;
2. The pathological biopsy was consistent with mantle cell lymphoma;
3. Measurable lesions on cross-sectional imaging recorded by diagnostic imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) (defined as the presence of at least one two-dimensional measurable lesion with a maximum cross-sectional diameter (GTD) ≥1.5 cm, regardless of the short axis diameter);
4. The physical status of the Eastern United States Cooperative Oncology Group (ECOG) ≤2 points;
5. Full liver function: upper limit of bilirubin≤3×normal value (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; Alkaline phosphatase (ALP) ≤5×ULN; Serum creatinine ≤1.5×ULN, or creatinine clearance rate calculated according to Cockcroft-Gault formula ≥35mL/min;
6. Voluntary participation, willingness to provide the above treatment data, signed and dated informed consent.

Exclusion Criteria:

1. Other clinical trials have been included;
2. Immunosuppressive therapy is being used for other diseases;
3. Lymphoma has been treated with other regimens before entry;
4. Complicated with other malignant tumors;
5. Those who are judged by the investigator to be unsuitable to participate in this study;
6. Serious mental or neurological disorder that affects informed consent and/or the presentation or observation of adverse reactions;
7. Patients who could not be followed up;

Exit (drop-off) criteria :

1. Subject requires to quit;
2. Serious adverse events occurred during the trial, so it is inappropriate to continue the clinical trial;
3. If the disease progresses during the study, it is inappropriate to continue using the experimental drug and/or cannot continue the study protocol;
4. Incomplete research data records;
5. Patients could not be followed up.Withdrawal cases should be retained for future reference and transferred from the last record to the final record for ITT analysis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with primary mantle cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
the overall response (complete response + partial response) | From the date of first study drug administration until the end of Cycle 2 (each cycle is 28 days)
  Objective response rate，sum of complete response rate and partial response rate of ibrutinib combination therapy in initial treatment of MCL
the overall response (complete response + partial response) | From the date of first study drug administration until the end of Cycle 6 (each cycle is 28 days)
  Objective response rate，sum of complete response rate and partial response rate of ibrutinib combination therapy in initial treatment of MCL

SECONDARY OUTCOMES:
Progression-free survival (PFS),OS,CR,DOR | 2 years
  Efficacy and survival of ibrutinib combination therapy in primary MCL, including: PFS,OS,CR,DOR
Incidence and severity of adverse events(AE) | 2 years
  Incidence of toxicity, defined as grade 3 or higher non-hematologic toxicity, grade 3 neutropenia, grade 4 hematologic toxicity, inability to administer full schedule and dose, or inability to receive treatment day 1 of course 2
The recurrence rate of MCL after initial treatment with ibrutinib | 2 years
  The recurrence rate of MCL after initial treatment with ibrutinib
Minimal residual disease negative (MRD-) rate of patients combination therapy | 1 year and 2 years
  MRD- rate will be estimated as the percentage of patients who achieved MRD-(ctDNA from Peripheral blood determined by NGS).

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, Professor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China